CLINICAL TRIAL: NCT01104766
Title: A Double-Blind, Placebo and Active-Controlled Evaluation of the Safety and Efficacy of Cariprazine in the Acute Exacerbation of Schizophrenia
Brief Title: Safety and Efficacy of Cariprazine in Patients With Schizophrenia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Forest Laboratories (Industry)
Collaborators: Gedeon Richter Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RGH-MD-04
Record Dates: First submitted 2010-04-09; First posted 2010-04-15 (Estimated); Results first posted 2018-10-29 (Actual); Last update posted 2018-10-29 (Actual); Status verified 2018-10

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Acute Schizophrenia; Psychotropic Drugs; Aripiprazole; Antipsychotic Agents; Mental Disorders; Dopamine Agents; Central Nervous System Agents
MeSH Terms: conditions — Schizophrenia; Mental Disorders | interventions — cariprazine; Aripiprazole

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Cariprazine 3mg (Experimental): Patients who meet eligibility criteria will be administered a once daily oral dose of cariprazine for six weeks. Upon completion of the study or early termination, patients will undergo a two week safety follow-up period.
  Interventions: Drug: Cariprazine
- Cariprazine 6mg (Experimental): Patients who meet eligibility criteria will be administered a once daily oral dose of cariprazine for six weeks. Upon completion of the study or early termination, patients will undergo a two week safety follow-up period.
  Interventions: Drug: Cariprazine
- Aripiprazole 10mg (Active Comparator): Patients who meet eligibility criteria will be administered a once daily oral dose of aripiprazole for six weeks. Upon completion of the study or early termination, patients will undergo a two week safety follow-up period.
  Interventions: Drug: Aripiprazole
- Placebo (Placebo Comparator): Patients who meet eligibility criteria will be administered a once daily oral dose of placebo for six weeks. Upon completion of the study or early termination, patients will undergo a two week safety follow-up period.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cariprazine — Patients who meet eligibility criteria will be administered a once daily oral dose of cariprazine for six weeks. Upon completion of the study or early termination, patients will undergo a two week safety follow-up period.
  Other Names: RGH-188
  Arms: Cariprazine 3mg; Cariprazine 6mg
Drug: Aripiprazole — Patients who meet eligibility criteria will be administered a once daily oral dose of aripiprazole for six weeks. Upon completion of the study or early termination, patients will undergo a two week safety follow-up period.
  Arms: Aripiprazole 10mg
Drug: Placebo — Patients who meet eligibility criteria will be administered a once daily oral dose of placebo for six weeks. Upon completion of the study or early termination, patients will undergo a two week safety follow-up period.
  Arms: Placebo

SUMMARY:
The objective of this study is to evaluate the efficacy, safety, and tolerability of cariprazine relative to placebo for the treatment of acute exacerbation of schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have provided informed consent prior to any study specific procedures
* Patients currently meeting the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition, Text Revision (DSM-IV-TR) criteria for schizophrenia (paranoid type, disorganized type, catatonic type or undifferentiated type), as confirmed by the Structured Clinical Interview for Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (SCID)
* Patients with normal physical examination, laboratory, vital signs,and/ or electrocardiogram (ECG)
* Current psychotic episode (schizophrenia exacerbation) < 2 weeks duration at Visit 1
* Structured Clinical Interview for the Positive and Negative Syndrome Scale (SCIPANSS) total score ≥ 80 and ≤ 120
* CGI-S score ≥ 4

Exclusion Criteria:

* Schizoaffective disorder, schizophreniform disorder, and other psychotic disorders
* Bipolar I and II disorder
* Pervasive developmental disorder, mental retardation, delirium, dementia, amnestic and other cognitive disorders
* DSM-IV-TR axis II disorder of sufficient severity to interfere with participation in this study
* Women who are pregnant or breast feeding

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 617 (Actual)
Dates: Start 2010-04-23 (Actual); Primary Completion 2011-12-20 (Actual); Study Completion 2011-12-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raffaele Migliore, MA, Study Director — Forest Laboratories
Locations (58):
- United States (20):
  - Woodland International Research Group, Inc., Little Rock, Arkansas
  - Woodland Research Northwest, LLC, Springdale, Arkansas
  - Synergy Clinical Research of Escondido, Escondido, California
  - Excell Research, Inc, Oceanside, California
  - Clinical Innovations, Inc., Riverside, California
  - Sharp Mesa Vista Hospital, San Diego, California
  - Collaborative Neuroscience Network, Inc., Torrance, California
  - Colorado Clinical Trials, Inc., Littleton, Colorado
  - Comprehensive Clinical Development, Inc., Washington D.C., District of Columbia
  - Florida Clinical Research Center, LLC, Bradenton, Florida
  - Hawaii Clinical Research Center, Honolulu, Hawaii
  - Uptown Research Institute, LLC, Chicago, Illinois
  - Alexian Brothers Center for Psychiatric Research, Hoffman Estates, Illinois
  - Precise Research Centers, Flowood, Mississippi
  - Millennium Psychiatric Associates, LLC, Creve Coeur, Missouri
  - CRI Worldwide, LLC, Willingboro, New Jersey
  - Windsor-Laurelwood Center for Behavioral Medicine, Willoughby, Ohio
  - Vanderbilt Psychiatric Hospital, Nashville, Tennessee
  - Claghorn-Lesem Research Clinic, Ltd., Houston, Texas
  - Pacific Institute of Medical Sciences, Bothell, Washington
- Romania (12):
  - Spitalul Clinic de Psihiatrie "Prof. Dr. Alexandru Obregia", Clinica X Psihiatrie, Bucharest
  - Spitalul Clinic de Psihiatrie 'Prof. Dr. Alexandru Obregia', Clinica III Psihiatrie, Bucharest
  - Spitalul Clinic de Psihiatrie 'Prof. Dr. Alexandru Obregia', Clinica VIII Psihiatrie, Bucharest
  - Spitalul Clinic Judetean de Urgenta Cluj, Clinica de Psihiatrie III, Cluj-Napoca
  - Spitalul Clinic de Neuropsihiatrie Craiova, Clinica II Psihiatrie, Craiova
  - Spitalul Clinic Militar de Urgenta, 'Dr. Stefan Odobleja' Clinical de Psihiatrie, Craiova
  - Spitalul Judetean de Urgenta Piatra Neamt, Piatra Neamţ
  - Spitalul Judetean de Urgenta Pitesti, Clinica de Psihiatrie, Piteşti
  - Spitalul de Psihiatrie Dr. Gheorghe Preda" Sibiu, Sibiu
  - Spitalul Judetean de Urgenta Targoviste, Sectia Psihiatrie, Târgovişte
  - Spitalul Clinic Judetean Mures, Clinica Psihiatrie I, Târgu Mureş
  - Spitalul Clinic Judetean de Urgenta Timisoara, Sectia Clinica de Psihiatrie "eduard Pamfil", Timișoara
- Russia (14):
  - Healthcare Institution "Moscow Regional Mental Hospital #5", Orekhovo-Zuyevo, Moscow Oblast
  - State Healthcare Institution <Arkhangelsk Regional Clinical Psychiatric Hospital>, Arkhangelsk
  - State Healthcare Institution "Regional Clinical Specialized Psychoneurological Hospital #1", Chelyabinsk
  - State Educational Institution of High Professional Education "Chita State Medical Academy of Roszdrav", Chita
  - St. Petersburg State Healthcare Institution "Mental Hospital #1 named after P.P Kashchenko", Gatchina
  - St. Petersburg State Healthcare Institution "St. Nicholas the Wonderworker Mental Hospital", Saint Petersburg
  - Federal State Budget Institution "St. Petersburg scientific-research psychoneurological Institute named after V.M Bekhterev" of the Ministry of Health and Social Development of the Russian Federation, Department of biological therapy of mental patients, Saint Petersburg
  - State institution "St. Petersburg scientifis-research psychoneurologic Institute of RosZdrav named after V.M Bekhterev", Saint Petersburg
  - Federal State Budget Institution "St. Petersburg scientific-research psychoneurological Institute named after V.M Bekhterev" of the Minitstry of Health and Social Development of the Russian Federation, Saint Petersburg
  - St. Petersburg State Healthcare Institution "City Mental Hospital #6 (hospital and Dispensary)", Saint Petersburg
  - St. Petersburg State Healthcare Institution "City Mental Hospital #3 named after I.I Skvortsov-Stepanov", department #7, Saint Petersburg
  - Municipal Healthcare Institution "City Clinical Hospital #2 named after V.I Razumovsky", Saratov
  - State Healthcare Institution "Saratov Saint Sophia Regional Mental Hospital", Saratov
  - Regional State Healthcare Institution "Tomsk Clinical Mental Hospital", Tomsk
- Ukraine (12):
  - Communal Institution of Kyiv Regional Council: Regional Psychiatric-Narcological Medical Association, Department #2 and #14, Village Glevakha, Kyiv Oblast
  - I.I. Mecnikov Regional Clinical Hospital, Regional Center of Psychosomatic Pathology, Dnipropetrovsk
  - Ukraine State Scientific and Research Institute of Medical and Social Problems of Disabiolity, Department of Psychoneurology, Psychotherapy and Medical Psychology, Dnipropetrovsk
  - Regional Clinical Psychiatric Hospital Department #11, M. Gorkyy Donetsk National Medical University, Chair of Psychiatry and Medical Psychology, Donetsk
  - Kharkiv Regional Clinical Psychiatric Hospital #3, Department #4, Department #14, Kharkiv
  - State Institution: Institute of Neurology, Psychiatry and Narcology of the AMS of Ukraine, Department of Borderline Psychic Pathology, Kharkiv
  - Kherson Regional Psychiatric Hospital, Department #3, Kherson
  - Kyiv City Clinical Psychoneurological Hospital #1, Center of Novel Treatment Methods and Rehabilitation of Psychotic Conditions, Kyiv
  - Communal Institution: Lviv Regional Clinical Psychiatric Hospital, Department #3 (male), Department #10 (female), Lviv
  - O.F. Maltsev Poltava Regional Clinical Psychiatric Hopspital, Department #3B, State Institution of Higher Education of Ukraine: Ukranian Medical Stomatological Academy, Chair of Psychiatry, Narcology and Medical Psychology, Poltava
  - Crimean Republican Institution: Clinical Psychiatric Hospital #1, Female Psychiatric Department #2, Male Psychiatric Department #1, S.I. Georgiyevskyy Crimean State Medical University, Chair of Psychiatry, Psychotherapy and Narcology, Simferopol
  - O.I. Yuschenko Vinnytsya Regional Psychoneurological Hospital, Department #10, Department #14, M.I. Pyrogov Vinnytsya National Medical University, Chair of Psychiatry and Narcology, Vinnytsia

REFERENCES:
- [Background] Citrome L, Durgam S, Lu K, Ferguson P, Laszlovszky I. The effect of cariprazine on hostility associated with schizophrenia: post hoc analyses from 3 randomized controlled trials. J Clin Psychiatry. 2016 Jan;77(1):109-15. doi: 10.4088/JCP.15m10192. PMID 26845266
- [Background] Earley W, Durgam S, Lu K, Laszlovszky I, Debelle M, Kane JM. Safety and tolerability of cariprazine in patients with acute exacerbation of schizophrenia: a pooled analysis of four phase II/III randomized, double-blind, placebo-controlled studies. Int Clin Psychopharmacol. 2017 Nov;32(6):319-328. doi: 10.1097/YIC.0000000000000187. PMID 28692485
- [Background] Nasrallah HA, Earley W, Cutler AJ, Wang Y, Lu K, Laszlovszky I, Nemeth G, Durgam S. The safety and tolerability of cariprazine in long-term treatment of schizophrenia: a post hoc pooled analysis. BMC Psychiatry. 2017 Aug 24;17(1):305. doi: 10.1186/s12888-017-1459-z. PMID 28836957
- [Result] Durgam S, Cutler AJ, Lu K, Migliore R, Ruth A, Laszlovszky I, Nemeth G, Meltzer HY. Cariprazine in acute exacerbation of schizophrenia: a fixed-dose, phase 3, randomized, double-blind, placebo- and active-controlled trial. J Clin Psychiatry. 2015 Dec;76(12):e1574-82. doi: 10.4088/JCP.15m09997. PMID 26717533
- [Derived] Laszlovszky I, Barabassy A, Nemeth G. Cariprazine, A Broad-Spectrum Antipsychotic for the Treatment of Schizophrenia: Pharmacology, Efficacy, and Safety. Adv Ther. 2021 Jul;38(7):3652-3673. doi: 10.1007/s12325-021-01797-5. Epub 2021 Jun 6. PMID 34091867
- [Derived] Barabassy A, Sebe B, Acsai K, Laszlovszky I, Szatmari B, Earley WR, Nemeth G. Safety and Tolerability of Cariprazine in Patients with Schizophrenia: A Pooled Analysis of Eight Phase II/III Studies. Neuropsychiatr Dis Treat. 2021 Apr 7;17:957-970. doi: 10.2147/NDT.S301225. eCollection 2021. PMID 33854317
- [Derived] Marder S, Fleischhacker WW, Earley W, Lu K, Zhong Y, Nemeth G, Laszlovszky I, Szalai E, Durgam S. Efficacy of cariprazine across symptom domains in patients with acute exacerbation of schizophrenia: Pooled analyses from 3 phase II/III studies. Eur Neuropsychopharmacol. 2019 Jan;29(1):127-136. doi: 10.1016/j.euroneuro.2018.10.008. Epub 2018 Nov 20. PMID 30470662
- [Derived] Cutler AJ, Durgam S, Wang Y, Migliore R, Lu K, Laszlovszky I, Nemeth G. Evaluation of the long-term safety and tolerability of cariprazine in patients with schizophrenia: results from a 1-year open-label study. CNS Spectr. 2018 Feb;23(1):39-50. doi: 10.1017/S1092852917000220. Epub 2017 May 8. PMID 28478771

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Randomization and treatment assignment were based on a randomization scheme prepared by Allergan Biostatistics prior to the start of the study. No-drug washout period of up to 7 days.
Groups:
- Placebo; Cariprazine 3.0 mg; Cariprazine 6.0mg; Aripiprazole 10.0 mg: Oral administration. Once per day.
Period: Overall Study
Arm/Group | Placebo | Cariprazine 3.0 mg | Cariprazine 6.0mg | Aripiprazole 10.0 mg
Started | 153 | 155 | 157 | 152
Completed | 95 | 104 | 97 | 114
Not Completed | 58 | 51 | 60 | 38
Not completed — Did not meet inc/exc criteria | 1 | 0 | 0 | 0
Not completed — Adverse Event | 17 | 15 | 20 | 14
Not completed — Lack of Efficacy | 20 | 15 | 14 | 8
Not completed — Protocol Violation | 2 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 17 | 19 | 25 | 15
Not completed — Lost to Follow-up | 1 | 2 | 1 | 1

BASELINE CHARACTERISTICS:
Population: The randomized population is also the safety population.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Cariprazine 3.0 mg | Cariprazine 6.0mg | Aripiprazole 10.0 mg | Total
Number analyzed (Participants) | 153 | 155 | 157 | 152 | 617
Age, Continuous [Mean (Standard Deviation); unit: Years] | 38.2 (11.3) | 37.9 (10.6) | 38.6 (10.6) | 39.3 (10.8) | 38.5 (10.8)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 97 | 99 | 100 | 94 | 390
  Female | 56 | 56 | 57 | 58 | 227
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 5 | 2 | 12
  Not Hispanic or Latino | 137 | 134 | 133 | 134 | 538
  Unknown or Not Reported | 13 | 19 | 19 | 16 | 67
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 93 | 102 | 101 | 99 | 395
  Black or African-American | 42 | 32 | 36 | 33 | 143
  Asian | 1 | 1 | 0 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 3 | 1 | 0 | 1 | 5
  Other | 2 | 2 | 3 | 1 | 8
  Missing | 12 | 17 | 17 | 16 | 62

OUTCOME MEASURES:

1. Primary Outcome: Measurement of Schizophrenia Symptoms: Change From Baseline in Positive and Negative Syndrome Scale (PANSS) Total Score.
Description: The Positive and Negative Syndrome Scale is a 30-item rating scale specifically developed to asses both the positive and negative symptom syndromes of patients with schizophrenia. The PANSS total score is rated based on a structured clinical interview with the patient and supporting clinical information obtained from family, hospital staff, or other reliable informants. This assessment provides scores in 9 clinical domains, including a positive syndrome, a negative syndrome, depression, a composite index, and general psychopathology. Each item is scored on a 7-point (1 to 7) scale, with 1 being minimal impact, and 7 being highest impact. The cumulative score ranges from 30 to 210. A negative change from baseline score indicates improvement.
Time Frame: Baseline to Week 6
Population: Intent-to-Treat Population, consisting of all patients in the Safety Population who had at least one postbaseline assessment of the PANSS total score.
Measure: Least Squares Mean (Standard Error); unit: Units on a Scale
Arm/Group | Placebo | Cariprazine 3.0 mg | Cariprazine 6.0mg | Aripiprazole 10.0 mg
Number analyzed (Participants) | 149 | 151 | 154 | 150
Units on a Scale | -14.3 (1.5) | -20.2 (1.5) | -23.0 (1.5) | -21.2 (1.4)
Statistical Analysis 1: Comparison: Placebo vs Cariprazine 3.0 mg; Test type: Superiority; p = 0.0044, ANCOVA; Mean Difference (Final Values) = -6.0, 95% CI 2-sided [-10.1 to -1.9]
Statistical Analysis 2: Comparison: Placebo vs Cariprazine 6.0mg; Test type: Superiority; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -8.8, 95% CI 2-sided [-12.9 to -4.7]
Statistical Analysis 3: Comparison: Placebo vs Aripiprazole 10.0 mg; Test type: Superiority; p = 0.0008, ANCOVA; Median Difference (Final Values) = -7.0, 95% CI 2-sided [-11.0 to -2.9]

2. Secondary Outcome: Measurement of the Overall Severity of Illness: Change From Baseline in Clinical Global Impression-Severity (CGI-S)
Description: The Clinical Global Impressions-Severity scale is a clinician-rated scale that measures the overall severity of a participant's illness in comparison with the severity of illness in other participants the physician has observed. The participant is rated on a scale from 1 to 7 with 1 indicating a "normal state" and 7 indicating "among the most extremely ill participants." A higher score indicates greater illness. A negative change from baseline score indicates improvement.
Time Frame: Baseline to Week 6
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Units on a Scale
Arm/Group | Placebo | Cariprazine 3.0 mg | Cariprazine 6.0mg | Aripiprazole 10.0 mg
Number analyzed (Participants) | 149 | 151 | 154 | 150
Units on a Scale | -1.0 (0.1) | -1.4 (0.1) | -1.5 (0.1) | -1.4 (0.1)
Statistical Analysis 1: Comparison: Placebo vs Cariprazine 3.0 mg; Test type: Superiority; p = 0.0004, ANCOVA; Mean Difference (Final Values) = -0.4, 95% CI 2-sided [-0.6 to -0.2]
Statistical Analysis 2: Comparison: Placebo vs Cariprazine 6.0mg; Test type: Superiority; p < 0.0001, ANCOVA; Median Difference (Final Values) = -0.5, 95% CI 2-sided [-0.7 to -0.3]
Statistical Analysis 3: Comparison: Placebo vs Aripiprazole 10.0 mg; Test type: Superiority; p = 0.0001, ANCOVA; Median Difference (Final Values) = -0.4, 95% CI 2-sided [-0.6 to -0.2]

ADVERSE EVENTS:
Time Frame: Assessed over 2 months
Description: Data is for the Double-blinding treatment period
Arm/Group | Placebo | Cariprazine 3.0 mg | Cariprazine 6.0mg | Aripiprazole 10.0 mg
All-Cause Mortality (participants affected / at risk) | 0/153 | 0/155 | 2/157 | 0/152
Serious Adverse Events (participants affected / at risk) | 2/153 | 4/155 | 7/157 | 4/152
Other Adverse Events (participants affected / at risk) | 68/153 | 61/155 | 71/157 | 61/152
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=153) | Cariprazine 3.0 mg (N=155) | Cariprazine 6.0mg (N=157) | Aripiprazole 10.0 mg (N=152)
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 1 | 0
Schizophrenia, paranoid type (Psychiatric disorders) | 0 | 1 | 1 | 0
Agitation (Psychiatric disorders) | 0 | 0 | 1 | 0
Complete Suicide (Psychiatric disorders) | 0 | 0 | 1 | 0
Dehydration (Renal and urinary disorders) | 0 | 0 | 1 | 0
Ischemic stroke (Cardiac disorders) | 0 | 0 | 1 | 0
Social stay hospitalization (Surgical and medical procedures) | 0 | 0 | 1 | 1
Transient ischemic attack (Nervous system disorders) | 0 | 0 | 1 | 0
Psychotic disorder (Psychiatric disorders) | 0 | 2 | 0 | 0
Schizophrenia (Psychiatric disorders) | 0 | 1 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0
Artropod bite (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 0 | 0 | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Placebo (N=153) | Cariprazine 3.0 mg (N=155) | Cariprazine 6.0mg (N=157) | Aripiprazole 10.0 mg (N=152)
Abdominal discomfort (Gastrointestinal disorders) | 3 | 1 | 7 | 9
Nausea (Gastrointestinal disorders) | 5 | 3 | 5 | 11
Vaginal Infection (Infections and infestations) | 0/56 | 3/56 | 0/57 | 0/58
Akathisia (Nervous system disorders) | 9 | 12 | 24 | 11
Headache (Nervous system disorders) | 17 | 10 | 16 | 15
Insomnia (Psychiatric disorders) | 25 | 21 | 22 | 16
Anxiety (Psychiatric disorders) | 11 | 12 | 12 | 12
Agitation (Psychiatric disorders) | 12 | 3 | 4 | 8
Schizophrenia (Psychiatric disorders) | 12 | 3 | 4 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All data generated in this study will be the property of Forest Research Institute, Inc. An integrated clinical and statistical report will be prepared at the completion of the study. Publication of the results by the Investigator will be subject to mutual agreement between the Investigator and Forest Research Institute, Inc.